CLINICAL TRIAL: NCT02226991
Title: A Single-centre, Open-label Study to Assess the Effects of Steady-state Efavirenz 600 mg QD (Sustiva®) on Tipranavir Concentration When Tipranavir/Ritonavir Are Administered at Doses 500 mg/200 mg BID to Steady-state in Healthy Adult Volunteers
Brief Title: Effects of Steady-state Efavirenz 600 mg QD (Sustiva®) on Tipranavir Concentration at Steady-state in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.102
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; efavirenz

ARMS (1):
- TPV/RTV/EFV (Experimental): tipranavir (TPV) + ritonavir (RTV) from day 1 to day 24 efavirenz (EFV) from day 10 to day 23
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Efavirenz

INTERVENTIONS:
Drug: Tipranavir
Drug: Ritonavir
Drug: Efavirenz

SUMMARY:
Study to investigate the effects of steady-state Efavirenz (600 mg QD) on the steady-state pharmacokinetics of Tipranavir (500 mg BID) coadministered with Ritonavir (200 mg BID)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 60 years of age inclusive
2. A Body Mass Index (BMI) between 18 and 29.9 kg/m2
3. Signed informed consent prior to trial participation
4. Ability to swallow multiple large capsules without difficulty
5. Acceptable laboratory values that indicate adequate baseline organ function at screening visit

   * Laboratory values are considered to be acceptable if the severity of any parameter is ≤Grade 1, based on the Division of AIDS (DAIDS)/AIDS Clinical Trials Group (ACTG) Grading Scale
   * All abnormal laboratory values >Grade 1 are subject to approval by the BI trial clinical monitor
6. Acceptable medical history, physical examination, and 12-lead ECG at screening
7. Willingness to abstain from the following starting 2 weeks prior to administration of any study medication and up until the end of the study:

   * Grapefruit or grapefruit juice, red wine, Seville oranges, St. John's Wort, and Milk Thistle
8. Willingness to abstain from alcohol starting 3 days prior to administration of any study medication up to the end of the study
9. Willingness to abstain from the following starting 3 days prior to pharmacokinetic (PK) sampling:

   * Garlic supplements and methylxanthine containing foods or drinks (including coffee, tea, cola, energy drinks, chocolate, etc.), apples or apple juice
10. Willingness to abstain from over-the-counter herbal medications for the duration of the study
11. Must be a non-smoker
12. Willingness to abstain from vigorous physical exercise during intensive PK days; Days 10 and 24
13. Reasonable probability for completion of the study

Exclusion Criteria:

1. Female subjects of reproductive potential who:

   * Have positive serum pregnancy test
   * Have not been using a barrier method of contraception for at least 3 months prior to participation in the study
   * Are not willing to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and 60 days after completion/termination of the trial
   * Are breast-feeding.
2. Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month prior to Day 1 and for the duration of the study.

   Due to long half-life, subjects using Depo-Provera® within six months prior to Day 1 will be excluded from participation in this study
3. Use of hormone replacement therapy within 1 month prior to Day 1 and anytime during the study
4. Participation in another trial with an investigational medicine within 2 months prior to Day 1 of this study
5. Use of any medication listed in Appendix 10.5 within 30 days prior to Day 1 of this study
6. Administration of antibiotics within 15 days prior to Day 1 and anytime during the study
7. History of acute illness within 60 days prior to Day 1

   * Subjects will be excluded for acute illnesses that occurred more than 60 days prior to Day 1 if, in the opinion of the investigator, the subject does not qualify as a healthy volunteer
8. Have serological evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV)
9. Have serological evidence of exposure to HIV
10. Alcohol or substance abuse within 1 year prior to screening or during the study
11. Blood or plasma donations within 30 days prior to Day 1 or during the study
12. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering TPV, RTV or EFV to the subject
13. History of a psychiatric disorder that required pharmacological or other psychological treatment
14. Subjects who have taken (within 7 days prior to Day 1) any over-the-counter or prescription medication that, in the opinion of the investigator in consultation with the sponsor's clinical monitor, might interfere with absorption, distribution, or metabolism of the study medications
15. Known hypersensitivity to sulphonamide class of drugs
16. Known hypersensitivity to TPV, RTV, EFV or antiretroviral drugs (marketed or experimental use as part of clinical research studies)
17. Known elevated liver enzymes in past trials with any compound
18. Inability to adhere to the protocol
19. Cautions or warnings in the RTV and EFV package insert which, in the opinion of the investigator, constitute grounds for subject exclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration at steady state (Cmax) | up to 12 hours after drug administration
Drug concentration in plasma at 12 hours after administration (Cp12h) | up to 12 hours after drug administration
  Tipranavir (TPV)
Last measured drug concentration in plasma (Cplast) | up to 12 hours after drug administration
  Ritonavir (RTV)
Area under plasma concentration time curve from 0-12 hours (AUC0-12h) | up to 12 hours after drug administration

SECONDARY OUTCOMES:
Trough plasma concentration (Cmin) | before drug administration
Time from dosing to the maximum concentration (tmax) | up to 12 hours after drug administration
Elimination half-life (t1/2) | up to 12 hours after drug administration
Oral clearance (CL/F) | up to 12 hours after drug administration
Volume of distribution (Vz/F) | up to 12 hours after drug administration
Number of subjects with adverse events | up to 38 days after first drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 38 days after first drug administration